CLINICAL TRIAL: NCT06689852
Title: MULTICENTRIC, RANDOMIZED, EVALUATOR BLINDED CLINICAL INVESTIGATION FOR THE EVALUATION OF EFFICACY AND SAFETY OF TWO PRODUCTS FOR THE TREATMENT OF ONYCHOMYCOSIS
Brief Title: CLINICAL INVESTIGATION FOR THE EVALUATION OF EFFICACY AND SAFETY OF TWO PRODUCTS FOR THE TREATMENT OF ONYCHOMYCOSIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23E1728
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-11

CONDITIONS: Onychomycosis
Keywords: onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary objective is to evaluate the effectiveness of Enriched and Loceryl® in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface compared to baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enriched (Experimental): To be used twice daily during 9 month
  Interventions: Device: Enriched
- Loceryl (Experimental): To be used 1 per week during 9 months
  Interventions: Drug: Loceryl 5%

INTERVENTIONS:
Device: Enriched — To be used twice a day
  Arms: Enriched
Drug: Loceryl 5% — To be used once a week
  Arms: Loceryl

SUMMARY:
The efficacy and safety of ENRICHED (X92001591) will be evaluated in a multicentric, randomized, evaluator blinded clinical investigation in 88 patients.

DETAILED DESCRIPTION:
Subjects will be treated with either the test medical device (ENRICHED X92001591) or the reference product (Loceryl, 5% amorolfine) for a period of 9 months. The primary objective of the investigation will be increase of % of healthy nail surface versus baseline, as evaluated by a blinded investigator. Subjects will be followed up for a period of 9 months, with visits at D0 (baseline), D90 (month 3), D180 (month 6) and D270 (month 9).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient having given freely her/his informed, written consent. 2. Patient having a good general health. 3. Age: between 18 and 70 years; 4. Patient with superficial onychomycosis on at least one great toenail or fingernail (for at least 10% in each arm) or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablets).

  5. Patient with positive KOH staining. 6. Patient cooperative and aware of the products modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.

  7. Patient being psychologically able to understand information and to give their/his/her consent.

  8. Patient having stopped any systemic antifungal treatment since at least 6 months before screening and/or any topical antifungal treatment since at least 3 months before screening.

  9. Patient who agree to refrain from receiving pedicure/manicure, artificial nails and/or cosmetic nail varnish or other medication on the nail being treated for the entire study duration.

  10. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after study end.

Exclusion Criteria:

- 1. Pregnant, breastfeeding woman or woman planning a pregnancy during the study; 2. Patient considered by the investigator likely to be non-compliant with the protocol. 3. Patient enrolled in another clinical trial or which exclusion period is not over. 4. Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk; 5. Patient suffering from a severe or progressive disease (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, HIV, psoriasis, lichen planus, immunosuppressive pathology… 6. Patient having a known allergy or hypersensitivity to one of the constituents of the tested products.

7. Patient with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Blinded evaluation of the percentage of healthy nail surface | 270 days
  Variation of the percentage of healthy surface after 270 days (9 months) of treatment with the test medical device or reference product versus baseline value. Blinded evaluation is done by digital analysis of photographs of the infected toenail or fingernail.

SECONDARY OUTCOMES:
Percentage of healthy surface (performance) | 90 days, 180 days
  Variation of the percentage of healthy surface after 90 days (3 months) and 180 days (6 months) of treatment with the test medical device or reference product versus baseline value. Blinded evaluation is done by digital analysis of photographs of the infected toenail or fingernail.
Mirobiological efficacy ; KOH staining (Performance) | 270 days
  Evaluation of microbiological efficacy of both treatments versus baseline by KOH staining and fungal culture at D270 (month 9)
Clinical efficacy: Visual appearance of nail (including onycholysis, nail dystrophy, nail discoloration and nail thickening) (Performance) | 90 days, 180 days, 270 days
  Assessment of clinical efficacy of both treatments on D0 (baseline), D90 (month 3), D180 (month 6) and D270 (month 9) by evaluation of the following parameters: onycholysis, nail dystrophy, nail discoloration, and nail thickening by the investigator in live.
  Each parameter is scored from 0 (none) - 4 (severe). The total score of all parameters is an indication of the visual appearance of the nail.
Clinical efficacy: onychomycosis evolution (Performance) | 90 days, 180 days, 270 days
  Assessment of onychomycosis evolution on D90 (month 3), D180 (month 6) and D270 (month 9) by the investigator in live
  * Failure: increase in the total infected area or aggravation
  * Status Quo
  * Improvement: decrease of the total infected area
  * Success: Disappearance of the total infected area
Impact on quality of life (Performance) | 180 days, 270 days
  Evaluation of the impact on the quality of life (QoL) of patients using a validated questionnaire (NailQoL) on D0 (baseline) and 180 (month 6) and 270 (month 9) days of treatment with the test medical device or reference, respectively
Subjective evaluation questionnaire for the patient (Performance) | 14 days, 90 days, 180 days, 270 days
  Evaluation of efficacy, tolerance, and acceptability of the test medical device and reference by thepatients using a subjective evaluation questionnaire, performed at D14, D90 (month 3), D180 (month 6) and D270 (month 9).
Evaluation of tolerance | 90 days, 180 days, 270 days
  Evaluation of tolerance of the test medical device and reference product at D90 (month 3), D180 (month 6) and D270 (month 9). Assessment is performed by the investigator via clinical evaluation and subject interrogation. The investigator will assign a score between 0 (bad tolerance) to 3 (very good tolerance).

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France, France

IPD SHARING:
Plan to Share IPD: No